CLINICAL TRIAL: NCT06642064
Title: Effects of Health Education on Physical Activity Promotion Based on PRECEDE-PROCEED Model Among Adolescents in Yunnan, China
Brief Title: Effects of Health Education on Physical Activity Promotion Based on PRECEDE-PROCEED Model Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Linxian (Other)
Responsible Party: Sponsor-Investigator, Zeng Linxian, Instructor, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: USM/JEPeM/22110706
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-08

CONDITIONS: Excessive Physical Exertion

STUDY DESIGN:
Intervention Model Description: Intervention group and Control group (2 groups):
  • Intervention group:
  Participants were invited to participate in a 20-minute interactive learning course (PPT lecture) and a 25-minute physical activity.The intervention lasted for 12 weeks, twice a week, 45 minutes each time, for a total of 1080 minutes.
  • Control group:
  Participants only received a logbook to record their physical activity every week and participated in regular physical exercise activities at school.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group and Control group (2 groups) (Experimental): This study held a group meeting before the formal experiment to guide all participants in advance and explain the entire experimental process to them in detail. Students with questions were given a unified and detailed explanation. Each participant received a health education manual and a physical activity record book. During the experimental stage, the researchers reminded the participants to attend the health education lectures and physical activity experiments on time. Participants were required to participate in the experiment according to the experimental content.
  Interventions: Behavioral: Intervention group
- control group (No Intervention): Control group: Participants only received a logbook to record their physical activity every week and participated in regular physical exercise activities at school

INTERVENTIONS:
Behavioral: Intervention group — • Intervention group:
  Participants were invited to participate in a 20-minute interactive learning course (PPT lecture) and a 25-minute physical activity.The intervention lasted for 12 weeks, twice a week, 45 minutes each time, for a total of 1080 minutes.
  Arms: Intervention group and Control group (2 groups)

SUMMARY:
A randomized controlled trial (RCT) was conducted to evaluate the changes in physical activity in adolescents before and after a health education program intervention based on the PRECEDE-PROCEED model.

DETAILED DESCRIPTION:
Based on the overall theoretical framework of the PRECEDE-PROCEED model, starting from the five steps of the PRECEDE-PROCEED model, namely, sociological evaluation, epidemiological evaluation, behavioral environment evaluation, educational organization evaluation, and management policy evaluation, a cross-sectional study was conducted to understand the physical activity level, vision, physical fitness level, social support, exercise self-efficacy, perceived benefits and barriers of exercise, and school sports environment support of adolescents of different genders and grades in Yunnan Province, China, and to analyze the paths of influencing factors. Based on the PRECEDE-PROCEED model, a health education program for promoting physical activity suitable for adolescents in Yunnan Province, China was developed, and an experimental intervention was conducted using a health education program based on the PRECEDE-PROCEED model. The effect of health education based on the PRECEDE-PROCEED model on promoting physical activity among adolescents in Yunnan Province was explored, so as to achieve the improvement of adolescent physical activity level and health promotion, and it is expected to provide a reference for the promotion of physical activity and physical health of adolescents in China.

Inclusion criteria:

* 15 to 18 years old, resident in Kunming, Yunnan, China;
* Adolescents who are understand the information that explained by the researcher and agree to be included in the study；
* Voluntarily participate in the experiment, cooperate with the research during the research process, and sign the informed consent；
* Adolescents who healthy to participate in physical activity (measured by PAR-Q).

Exclusion criteria:

* Mental illness with cognitive impairment;
* People with speech or ear dysfunction;
* Recent or upcoming surgery (within 3 months), or commonalities;
* Subjects During the research period, if symptoms of discomfort occur, they are asked to stop and withdraw according to the subject's own will;
* Have participated in similar research in the past. People who meet any of the exclusion criteria are not included in the study.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 18 years old, resident in Kunming, Yunnan, China;
* Adolescents who are understand the information that explained by the researcher and agree to be included in the study；
* Voluntarily participate in the experiment, cooperate with the research during the research process, and sign the informed consent；
* Adolescents who healthy to participate in physical activity (measured by PAR-Q).

Exclusion Criteria:

* Mental illness with cognitive impairment;
* People with speech or ear dysfunction;
* Recent or upcoming surgery (within 3 months), or commonalities;
* Subjects During the research period, if symptoms of discomfort occur, they are asked to stop and withdraw according to the subject's own will;
* Have participated in similar research in the past. People who meet any of the exclusion criteria are not included in the study.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 194 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Health education based on the PRECEDE-PROCEED model has a positive impact on promoting physical activity among adolescents in Yunnan Province | 12 weeks
  This study collected data via questionnaires, physical fitness tests, and vision assessments. Instruments included validated questionnaires-ASAFA-C, Q-SPACE-C, EBBS-CN, PAQ-CN, and S-PASESC-measuring social support, school environment, perceived benefits/barriers, activity levels, and self-efficacy. Physical tests per NSPFH 2014 included BMI, sprints, runs, jumps, pull-ups/sit-ups, and vital capacity. Data were analyzed using descriptive statistics and repeated measures ANOVA/MANOVA over four measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Linxian Zeng, PHD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Anning No. 1 Middle School in KunMing,Yunnan Province, China, Kunming, Yunnan, China